CLINICAL TRIAL: NCT02447224
Title: A Pilot Study for a Randomized Trial of Antibiotics Versus Surgery for Treatment of Patients With Acute Uncomplicated Appendicitis
Brief Title: Pilot Trial of Antibiotics Versus Surgery for Treating Acute Appendicitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Olive View-UCLA Education & Research Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, David A. Talan, Principal Investigator, Olive View-UCLA Education & Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R21DK102048 (NIH)
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Acute Uncomplicated Appendicitis
Keywords: appendicitis; non operative management; appendectomy
MeSH Terms: conditions — Appendicitis | interventions — Metronidazole; Appendectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotics (Experimental): Once-a-day dose of IV/IM ertapenem for at least two days and cefdinir and metronidazole, to complete 10 days total antibiotic therapy.
  Interventions: Drug: 1 gm IV ertapenem at enrollment; Drug: 1 gm IV ertapenem at Day 2 and oral metronidazole and cefdinir to complete 10 days
- Appendectomy (Active Comparator): Patients in the surgery therapy arm will only receive one dose of IV ertapenem prior to surgery.
  Interventions: Drug: 1 gm IV ertapenem at enrollment; Procedure: Appendectomy

INTERVENTIONS:
Drug: 1 gm IV ertapenem at enrollment
Drug: 1 gm IV ertapenem at Day 2 and oral metronidazole and cefdinir to complete 10 days
  Arms: Antibiotics
Procedure: Appendectomy
  Arms: Appendectomy

SUMMARY:
The major goal of the project is to demonstrate the feasibility of conducting a multi-center randomized clinical trial of antibiotic therapy versus appendectomy for the treatment of patients with acute uncomplicated appendicitis by conducting a single-site pilot study so as to optimize the chance of a large multi-center clinical trial's future success.

DETAILED DESCRIPTION:
This will be a single-site open clinical trial in which subjects with acute uncomplicated appendicitis are randomized to one of two initial treatment strategies, surgery with peri-operative antibiotics or antibiotics alone, with surgical rescue if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Adult or child ages ≥5 years;
* Diagnosis of acute uncomplicated appendicitis, confirmed by CT, ultrasound and/or MRI performed within 24 hours of consent, as read by an attending radiologist, and confirmed by consultation of an attending surgeon;
* Ability to provide written informed consent (and for subjects ages 5-17, consent from their parent/guardian and assent if applicable); and
* Negative pregnancy test for subjects who are women of childbearing potential.

Exclusion Criteria:

* instability/severe sepsis, appendiceal perforation by imaging, serious co-morbidities limiting randomization, pregnancy, and inability to complete the treatment protocol.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Major Complications | 30 days
  The American College of Surgeons (ACS) National Surgical Quality Improvement Program (NSQIP) criteria and definitions for major complications will be used. In addition, antibiotic related complications will be evaluated, i.e., antibiotic-related/Clostridium difficile colitis and antibiotic reaction requiring hospitalization.

SECONDARY OUTCOMES:
Recurrent appendicitis | 30 days
QOL outcomes | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Olive View-UCLA Medical Center, Sylmar, California, United States